CLINICAL TRIAL: NCT05999643
Title: Characterizing Spondyloarthritis With 68Ga-FAPI PET/CT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAPI in SpA
Record Dates: First submitted 2023-07-30; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-07

CONDITIONS: Spondyloarthritis; Axial Spondyloarthritis; Ankylosing Spondylitis
Keywords: Spondyloarthritis; Axial Spondyloarthritis; Ankylosing Spondylitis; 68Ga-FAPI
MeSH Terms: conditions — Spondylarthritis; Axial Spondyloarthritis; Spondylitis, Ankylosing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inject 68Ga-FAPI and then perform PET/CT scan. (Experimental): Inject 68Ga-FAPI and then perform PET/CT scan
  Interventions: Diagnostic Test: Drug: 68Ga-FAPI

INTERVENTIONS:
Diagnostic Test: Drug: 68Ga-FAPI — Intravenous injection of one dosage of 111-185 MBq (3-5 mCi) 68Ga-FAPI. Tracer doses of 68Ga-FAPI will be used to image SpA lesions in SI joints, spine, musculoskeletal and the extra-articular involvement by PET/CT.
  Other Names: 68Ga-fibroblast activating protein inhibitors

SUMMARY:
To evaluate the potential usefulness of 68Ga-FAPI PET/CT for the diagnosis, inflammation evaluation and prognosis prediction in spondyloarthritis.

DETAILED DESCRIPTION:
Spondyloarthritis (SpA) is a chronic inflammatory rheumatic disease characterized by inflammatory back pain, enthesitis, dactylitis, and the formation of syndesmophytes, all of which significantly affect a patient's healthy functioning and general quality of life. Prevalence of underlying malignancy is high in patients with SpA. Radiographic sacroiliitis became a crucial finding in the diagnosis and classification of patients.

68Ga-FAPI has been developed as tracers specific for fibroblast-activation protein (FAP), which is overexpressed in activated fibroblasts in various type of cancers and autoimmune diseases, such as rheumatoid arthritis, IgG4-related diseases and interstitial lung diseases.

Recently the investigators have published articles of the application of 68Ga-FAPI in IgG4-related disease and rheumatoid arthritis, which showed it was more sensitive than FDG in detecting a certain type of inflammation. Increased 68Ga-FAPI Uptake in ankylosing spondylitis in a patient with rectal cancer has also been reported in a case report, indicating the potential utility of FAP-targeted PET/CT imaging for diagnosis and disease assessment in spondyloarthritis.

Thus, this prospective study is going to investigate utility of 68Ga-FAPI PET/CT in diagnosis of spondyloarthritis as well as inflammation assessment in joints including the sacroiliac (SI) joints, spine and peripheral joints. Also, this study aims to investigate potential utility of 68Ga-FAPI PET/CT in predicting treatment response and disease prognosis such as formation of syndesmophytes and erosive changes.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of SpA according to the ASAS (Assessment of Spondyloarthritis International Society) classification criteria for SpA.
2. Adult men or women 18 and ≤ 65 years of age at the time of signing the informed consent (ICF).
3. participants who were able to provide informed consent (signed by participant or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

1. Pregnancy;
2. Breastfeeding;
3. known allergy against FAPI;
4. any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
To define the distribution pattern of 68Ga-FAPI in SpA patients. | 60 minutes following injection
  To quantify 68Ga-FAPI tracer biodistribution in characteristic inflammatory tissue including SI joints, spine, and the peripheral joints versus conventional x ray examination or magnetic resonance imaging (MRI) techniques in adult active SpA. 68Ga-FAPI PET tracer biodistribution will be assessed by semi-quantitative analysis (unit/metrics = standardized uptake values (SUV)).

SECONDARY OUTCOMES:
Correlation between uptake of 68GA-FAPI and other parameters associated with disease activity. | 30 days
  Correlation between uptake of 68GA-FAPI and parameters associated with disease activity including Ankylosing Spondylitis Disease Activity Score (ASDAS), Bath ankylosing spondylitis disease activity index (BSADAI）, Bath ankylosing spondylitis functional index (BASFI)，and Maastricht Ankylosing Spondylitis Enthesitis Score（MASES). The Standardized uptake value (SUV) of 68Ga-FAPI was calculated and analyzing the correlation between pathological results and parameters associated with disease activity.
Correlation between uptake of 68GA-FAPI change and disease activity change | Up to 2 years
  Correlation between change in standardized uptake value (SUV) of 68Ga-FAPI at inflammatory site with change in Ankylosing Spondylitis Disease Activity Score (ASDAS), Bath ankylosing spondylitis disease activity index (BSADAI), Bath ankylosing spondylitis functional index (BASFI)，and Maastricht Ankylosing Spondylitis Enthesitis Score（MASES) at different disease stage.
Correlation between uptake of 68GA-FAPI and therapy response | Up to 2 years
  Percentage of participants achieving ankylosing spondylitis disease activity score inactive disease [ASDAS ID (<1.3)] after 1 year standardized treatment in participants with high standardized uptake value (SUV) of 68Ga-FAPI and low standardized uptake value (SUV) of 68Ga-FAPI at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Guixiu Shi, PhD, Study Director — The First Affiliated Hospital of Xiamen University
Locations (1):
- The first affiliated hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen Y, Yu L, Chen S, Liu W, Han H, Pang Y, Lin Q, Li Y, Chen L, Cai J, Zhao L, Sun L, Shi G, Chen H, Liu Y. Fibroblast activation protein-targeted PET/CT with 68Ga-FAPI-46 for evaluation of structural damage and inflammation in axial spondyloarthritis: a prospective study. Eur J Nucl Med Mol Imaging. 2025 Oct;52(12):4661-4673. doi: 10.1007/s00259-025-07310-2. Epub 2025 May 1. PMID 40310563